CLINICAL TRIAL: NCT05932732
Title: A Phase IV Open-label Trial Assessing the Impact on Skin Quality, Hydration, and Barrier of Three (3) Hydrafacial Treatments in Adults of Fitzpatrick Skin Types I-VI
Brief Title: Trial Assessing the Impact on Facial Skin Quality, Hydration, and Skin Barrier of Three (3) Hydrafacial Treatments in Adults of All Skin Types.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Austin Institute for Clinical Research (Network)
Collaborators: The HydraFacial Company (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDCR-000300
Record Dates: First submitted 2023-06-15; First posted 2023-07-06 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-07

CONDITIONS: Cutis Laxa Facialis; Xeroderma
MeSH Terms: conditions — Ichthyosis

STUDY DESIGN:
Intervention Model Description: Approximately 5 subjects of each Fitzpatrick skin types I-VI will be included, with a total of 30 subjects participating, assessing efficacy and subject satisfaction, before and after three (3) hydrafacial treatments each performed 28 days apart.
Masking Description: Not applicable, no masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HydraFacial Syndeo Treatment (Other): Three HydraFacial Syndeo Treatment will be performed 28 days apart at the Pflugerville site.
  Interventions: Device: HydraFacial Syndeo System; Drug: ReGen-GF
- Hydrafacial Elite MD Treatment (Other): hree HydraFacial Elite MD Treatment will be performed 28 days apart at the Houston site.
  Interventions: Drug: ReGen-GF; Device: HydraFacial Elite MD System

INTERVENTIONS:
Device: HydraFacial Syndeo System — Utilizing patented Vortex Fusion Technology, a pneumatic device, the HydraFacial Syndeo system cleanses, exfoliates, and hydrates the skin.
  Arms: HydraFacial Syndeo Treatment
Drug: ReGen-GF — The Regen-GF Booster, a serum formulated to increase collagen and elastin production, will be used during each HydraFacial treatment using the HydraFacial handpiece and specialized tip for application. Ingredients include Heptapeptide-32 maintains the appearance of healthy, youthful skin through collagen and elastin production, Copper Peptide Cu-GHK regenerates healthy-looking skin by accelerating wound healing and skin repair, Palmitoyl Tetrapeptide-7 treats inflammation while boosting the growth of collagen-producing tissues, Palmitoyl Tripeptide-5 helps skin cells flush toxins while enhancing the appearance of firmness, Azelaoyl Bis-Dipeptide 10 addresses signs of aging by managing the formation of free radicals, K3 Vitamin C promotes collagen synthesis, and Hyaluronic Acid hydrates the skin.
Device: HydraFacial Elite MD System — Utilizing patented Vortex Fusion Technology, the HydraFacial Elite MD system cleanses, exfoliates, and hydrates the skin.
  Arms: Hydrafacial Elite MD Treatment

SUMMARY:
This is a phase IV, unblinded, open-label study assessing the impact on skin quality, hydration, and barrier of three (3) Hydrafacial treatments in healthy adults of Fitzpatrick Skin Types I & II, III, IV, V & VI, 30 to 55 years of age. Efficacy and subject satisfaction will be assessed, before and after three (3) HF treatments, in 6 patient cohorts, each cohort defined by FST I-VI.

DETAILED DESCRIPTION:
A multisite study. Approximately 30 subjects will be enrolled in the trail. The purpose of this study is to assess the changes in facial skin hydration and moisturization after a series of 3 hydrafacial treatments in subjects of all Fitzpatrick skin types. In addition, patient and investigator assessed changes in skin quality characteristics will be captured. The primary object is Improvement in skin quality assessments performed by the investigator from baseline (prior to treatment 1) to Day 85, the final study visit.

Utilizing patented Vortex Fusion Technology, a pneumatic device, the HydraFacial Syndeo system and HydraFacial Elite MD system cleanses, exfoliates, and hydrates the skin. The procedure lasts 30-45 minutes and includes three steps: a gentle cleansing, followed by a light peel and then infusion of a proprietary blend of ingredients, termed the Regen GF booster, which contains growth factors, humectants and moisturizers. Once this treatment is complete subjects will undergo a non-invasive red LED treatment, Ellipse Red Light, during which the skin is exposed to gentle red light under a horseshoe-shaped illumination device while wearing blocking goggles, to improve circulation and reduce inflammation.

The first visit, including screening and baseline with HF treatment #1, is followed by two additional HF treatments 28 days apart, with a final visit occurring on day 85. PROs, including satisfaction are captured, as well as Investigator-assessed measurements of skin quality (using the validated Scientific Assessment Scale of Skin Quality) including elasticity, roughness, fine lines, pigmentation, erythema, and pore size, Investigator Global Aesthetic Improvement Scale, and Investigator Tolerability Assessment. Additionally, corneometry (a measurement of skin hydration) and tewlometry (a measure of transepidermal water loss, assessing the integrity of the skin barrier) are performed to assess changes with the treatments at selected time points.

All adverse events observed by the study site personnel, or reported spontaneously by the subject, will be recorded, including description, assessment of severity, and relationship to study treatment. Study site will document all serious adverse events that occur (whether or not related to study treatment). The collection period for all SAEs will begin after informed consent is obtained and end after procedures for the final study visit have been completed. The site investigator will report SAEs in accordance with the standard operating procedures and policies of the local Institutional Review Board (IRB).

Subjects are free to withdraw from participating in this study at any time and for whatever reason, specified or unspecified, and without prejudice. Subjects who terminate early will be asked to complete, if possible, all assessments and procedures that would have been conducted on the last study visit.

It is the responsibility of the site investigator to identify and report deviations within 5 working days of identification of the protocol deviation. All deviations must be addressed in study source documents, reported to the study sponsor, and the reviewing Institutional Review Board (IRB) per their policies.

This is an exploratory study for which results will be reported, but not analyzed with statistical tools beyond calculating mean values. No interim analyses will be conducted. This study will use web-based, electronic case report forms (eCRFs) developed through a validated, Electronic Records/Electronic Signatures-compliant platform (US Title 21 CFR Part 11). The Investigator is responsible for all data entered via the remote data capture (RDC) system from the eCRFs and must confirm the accuracy of the data by electronically approving (signing) the eCRFs. The Sponsor will review the database to identify data errors or inconsistencies, which will be posted in the RDC system as queries for resolution.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females of Fitzpatrick skin types I-VI 30-55 years of age.
2. No known medical conditions that in the investigator's opinion may interfere with study participation.
3. Agrees to abstain from starting a new skincare product for the duration of trial participation.
4. Willingness to cooperate and participate by following study requirements.
5. Individuals must sign an informed consent and photography consent.

Exclusion Criteria:

1. History of any cancer excluding fully treated basal cell carcinoma or squamous cell carcinoma in situ in the treatment area.
2. Presence of untreated precancerous lesions in the treatment area.
3. Presence of sunburn, moderate to pronounced suntan, uneven skin tone, tattoos, scars or other disfiguration in the treatment area.
4. Any cutaneous condition that may affect study adherence or ability to assess endpoints, as determined by the investigator, to include, but not limited to, uncontrolled psoriasis, atopic dermatitis, severe photodamage, and uncontrolled acne.
5. Subject is pregnant, nursing, or planning to become pregnant.
6. Significant past medical history of hepatic, hypertensive, renal, cardiac, pulmonary, digestive, hematological, neurological, or psychiatric disease, which in the opinion of the Investigator would compromise the safety of the subject.
7. Currently participating in another clinical trial.
8. History of Photo Epilepsy.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-10-09 (Actual); Study Completion 2024-10-09 (Actual)

PRIMARY OUTCOMES:
Change in skin facial skin elasticity, wrinkles, roughness, fine lines, pigmentation, erythema, and pore size | Change from Baseline to Day 85
  Measured by Investigator assessment using the validated Scientific Assessment Scale of Skin Quality. the scale assesses the facial skin elasticity, wrinkles, roughness, fine lines, pigmentation, and erythema. The parameters include 0 = none (best possible outcome), 1 = mild, 2 = moderate, 3 = severe, and 4 = very severe (worst possible outcome). Pore size will be measured using parameters of 0 = fine (best possible outcome), 1 = small, 2 = moderate, 3 = large, and 4 = very large (worst possible outcome).
Change in facial aesthetic appearance | Change from Baseline to Day 85
  Measured by the Investigator Global Aesthetic Improvement Scale. Scale and parameters include 1 = worst (worst possible outcome), 2 = mildly improved, 3 = improved, 4 = much improved, and 5 = very much improved (best possible outcome).
Change in subjective irritation parameters | Change from Baseline to Day 85
  Measured by the Investigator Tolerability Assessment. Scale includes burning, stinging, and itching. Each will be measured by the following parameters, 0 = none (best possible outcome), 1 = mild, 2 = moderate, and 3 = severe (worst possible outcome).
Change in facial skin hydration | Change from Baseline to Day 85
  The Corneometry device will be used as a measurement of skin hydration. The values of skin hydration degree is between 0-130 arbitrary units (AU). The higher the value means a better outcome.
Change in transepidermal water loss | Change from Baseline to Day 85
  The Tewlometry device will be used as a measurement of transepidermal water loss. The units of measurement are grams of water per square meter per hour. The higher the value means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Lain, MD, MBA, Principal Investigator — Austin Institute for Clinical Research
Locations (2):
- United States (2):
  - Austin Institute for Clinical Research, Inc., Houston, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas